CLINICAL TRIAL: NCT02053558
Title: Tranversus Abdominis Plane (TAP) Block vs. Systemic Lidocaine to Improve Quality of Recovery After Outpatient Laparoscopic Surgery: A Non-inferiority, Randomized, Double Blinded, Placebo Controlled Trial
Brief Title: (TAP) Block vs. Systemic Lidocaine: Effects on Recovery
Acronym: TAP
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Could not obtain dedicated ultrasound device.
Sponsor: Northwestern University (Other)
Responsible Party: Principal Investigator, Meghan Rodes, Principal Investigator, Northwestern University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: STU00086849
Record Dates: First submitted 2014-01-30; First posted 2014-02-03 (Estimated); Last update posted 2019-12-16 (Actual); Status verified 2019-12

CONDITIONS: Pain; Surgery
Keywords: Anesthesiology; Pain; TAP block; Gynecology; Postoperative; Analgesia
MeSH Terms: conditions — Pain; Agnosia | interventions — Lidocaine; Ropivacaine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Systemic lidocaine (Placebo Comparator): Systemic lidocaine group will receive a lidocaine 1.5 mg/kg bolus after induction of anesthesia followed by a 2mg/kg/hr infusion and sham bilateral TAP blocks with normal saline 15mL on each side.
  Interventions: Drug: Systemic lidocaine
- TAP BLOCK with ropivacaine (Active Comparator): TAP block will receive bilateral TAP blocks using ultrasound guidance with 0.5% ropivacaine 15mL on each side and a bolus and infusion of normal saline after induction of anesthesia.
  Interventions: Drug: TAP BLOCK with ropivacaine

INTERVENTIONS:
Drug: Systemic lidocaine — Systemic lidocaine group will receive a lidocaine 1.5 mg/kg bolus after induction of anesthesia followed by a 2mg/kg/hr infusion and sham bilateral TAP blocks with normal saline 15mL on each side.
  Other Names: lidocaine 1 %
  Arms: Systemic lidocaine
Drug: TAP BLOCK with ropivacaine — TAP block group will receive bilateral TAP blocks using ultrasound guidance with 0.5% ropivacaine 15mL on each side and a bolus and infusion of normal saline after induction of anesthesia.
  Other Names: Ropivacaine .5%
  Arms: TAP BLOCK with ropivacaine

SUMMARY:
It has been demonstrated that female patients have poor quality of surgical recovery compared to male patients. Increased sensitivity to pain and increased susceptibility to postoperative nausea and vomiting have been attributed as causal factors. Currently, few strategies have been shown to improve quality of recovery in female patients undergoing laparoscopic hysterectomy. A better recovery in female patients undergoing outpatient laparoscopy is particularly desirable since those patients do not have access to potent intravenous medications and nursing support after hospital discharge.

Our group has previously demonstrated that both TAP block and systemic lidocaine improve quality of recovery after outpatient laparoscopic gynecological surgery. The TAP block, however, requires expertise, equipment (ultrasound), and additional time to perform as compared with a simple lidocaine infusion. It is currently unknown if a systemic lidocaine infusion provides non-inferior quality of recovery when compared to TAP block for outpatient laparoscopic gynecological surgery.

The main objective of the current investigation is to examine the effect of TAP block on quality of recovery compared to a systemic lidocaine infusion. We hypothesize that systemic lidocaine infusion would provide non-inferior quality of recovery when compared to TAP block for outpatient laparoscopic gynecological surgery.

Significance: This is the first study to compare systemic lidocaine to TAP block with regard to quality of recovery.

The research question; does systemic lidocaine provide similar quality of recovery as TAP block for outpatient laparoscopy? The hypothesis; systemic lidocaine provides non-inferior quality of recovery as TAP block for outpatient laparoscopy.

Research significance: It has been shown that females have poor surgical recovery compared to males; this project intends to demonstrate that systemic lidocaine provides similar recovery as TAP blocks but it does not require the expertise, equipment, and time needed to perform TAP blocks.

ELIGIBILITY:
Inclusion Criteria:

* Age: 18-65 years of age
* Surgery type: Outpatient Gynecological Laparoscopy
* ASA status: I and II
* Fluent in English

Exclusion Criteria:

* History of allergy to local anesthetics
* History of chronic opioid use
* Pregnant patients
* Drop Out: Conversion to open surgery, patient or surgeon request.

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2014-11-03 (Actual); Primary Completion 2017-02 (Actual); Study Completion 2017-02 (Actual)

PRIMARY OUTCOMES:
QoR-40 global score at 24 hours | 24 hours post operative
  QoR-40 global score at 24 hours

SECONDARY OUTCOMES:
Morphine consumption at 24 hours post operative | 24 hours post operative
  Total amount of morphine used in the 24 hour period post operative.

CONTACTS AND LOCATIONS:
Overall Officials: Meghan Rodes, MD, Principal Investigator — Northwestern University

IPD SHARING:
Plan to Share IPD: No